CLINICAL TRIAL: NCT03072550
Title: A Multi Center Open Label Early Feasibility Study to Evaluate the Efficacy and Safety of the RenewalNail™ Plasma Treatment System in Patients With Mild to Moderate Onychomycosis (Fungal Nail) of the Hallux Caused by Trichophyton Rubrum or Trichophyton Mentagrophytes.
Brief Title: Early Feasibility Study to Evaluate the Efficacy and Safety of the RenewalNail™ Plasma Treatment System in Patients With Mild to Moderate Onychomycosis (Fungal Nail)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DeviceFarm, Inc. (Industry)
Collaborators: Symbio, LLC (Industry); Center for Dermatology Clinical Research, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFCR-0002
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Results first posted 2019-08-29 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-08

CONDITIONS: Onychomycosis Due to Trichophyton Rubrum; Onychomycosis Due to Trichophyton Mentagrophytes
Keywords: fungal nail; toenail fungus

STUDY DESIGN:
Intervention Model Description: multi-center open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Multi-center open label (Experimental): Thirty Subjects with 20-75% Distal Subungual Onychomycosis (mild to moderate DSO) infection of their big toe (hallux) nail infected by the dermatophytes Trichophyton (T.) rubrum or T. mentagrophytes will be enrolled. All Subjects will receive three 45-minute plasma treatments performed over a week.
  Interventions: Device: RenewalNail™ Plasma Treatment System

INTERVENTIONS:
Device: RenewalNail™ Plasma Treatment System — application of cold atmospheric plasma to a fungal infected toenail
  Other Names: cold atmospheric plasma treatment

SUMMARY:
Early feasibility study to determine if a three-treatment protocol with the RenewalNail™ plasma treatment system over a week will result in mycological cure and/or clear nail growth on the treated hallux toe.

DETAILED DESCRIPTION:
The Sponsor has developed the RenewalNail™ plasma treatment system to topically treat fungal infected toenails. The goal of the RenewalNail™ therapy is to overcome the shortcomings of both topical and oral therapies by combining the safety of a topical treatment with the efficacy of an oral treatment.

The primary objective of this early feasibility study is to evaluate the efficacy and safety of the RenewalNail™ plasma treatment system and Protocol in achieving mycological cure for the patient. The Protocol calls for three 45-minute treatments performed over a week to achieve mycological cure. Mycological cure will be assessed with two consecutive mycological culture tests done over a week. Two consecutive negative results will confirm the elimination of fungus causing onychomycosis infection, as recommended by recent FDA guidance. There will be no placebo arm in the study.

Secondary objectives include assessing if the treatment protocol results in clear nail growth for the patient over a 5-month interval.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are between 21 to 75 years (inclusive) of age;
* Subjects male or female and of any race;
* Subjects who are in good general health and free from any clinically significant disease that might interfere with the study evaluations.
* Subjects with established clinical diagnosis of distal subungual onychomycosis;
* Subjects with at least one or both big toe nails involved with 20-75% infection;
* Subjects with both positive KOH and culture for onychomycosis dermatophytes in screening of nail samples;
* Subjects whose infection is confirmed to be caused by T. rubrum or T. mentagrophytes;
* Subjects who are willing and able to refrain from employing other (non-study) treatments (traditional or alternative) for his or her toenail onychomycosis throughout study participation;
* Subjects who are willing and able to refrain from the use of nail cosmetics such as clear and/or colored nail lacquers throughout study participation;
* Subjects who are willing and able to give written informed consent and able to adhere to procedures and visit schedules;
* Women of childbearing potential who are currently sexually active must agree to use a medically accepted method of contraception while receiving protocol specified treatment. Methods include condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed intrauterine device, oral or systemic hormonal contraceptive (plus an additional reliable barrier method), surgical sterilization (e.g., hysterectomy or tubal ligation);
* Women of childbearing potential who are not currently sexually active must agree to use a medically accepted method of contraception should they become sexually active while participating in the study;
* Women of childbearing potential must have a negative pregnancy test prior to start of study.

Exclusion Criteria:

* Subjects with presence of dermatophytoma (defined as demarcated and localized thick masses) of fungal hyphae and necrotic keratin between the nail plate and nail bed) on the target nail;
* Subjects with onychomycosis infection involving lunula of the affected toenail(s) or spikes of disease extending to nail matrix in the affected big toenail(s);
* Subjects with conditions other than distal subungual onychomycosis known to cause abnormal nail appearance such as psoriasis, severe moccasin-type tinea pedis requiring treatment, symptomatic interdigital tinea pedis, lichen planus, or other abnormalities that could result in a clinically abnormal nail;
* Subjects whose foot is too large (larger than US men's size 13) or too small (smaller than US women's size 3) to properly fit into the plasma treatment device;
* Subjects with a history of multiple repeated failures with previous therapies for onychomycosis;
* Subjects whose affected big toenails cannot become normal in the opinion of the investigator;
* Subjects with abnormality of the affected big toenail(s) that could prevent a normal appearing nail if clearing of infection is achieved;
* Subjects with trauma to the affected big toenail(s) as identified by the study doctor;
* Subjects who received topical antifungal treatment of the nails within 2 weeks before study initiation;
* Subjects who received systemic antifungal treatment within 3 months before study initiation;
* Subjects with dementia or psychic condition that might interfere with the ability to understand the study and thus give written informed consent;
* Simultaneous participation in another clinical study or participation in another clinical study in the 30 days directly preceding treatment;
* Subjects who are unwilling or unable to refrain from employing other (non-study) treatments (traditional and alternative) for their toenail onychomycosis throughout study participation;
* Subjects who are unwilling or unable to refrain from the use of nail cosmetics such as clear and/or colored nail lacquers until the end of study participation;
* Subjects who are immunocompromised (e.g. adrenal insufficiency, diabetes mellitus, febrile neutropenia, and the human immunodeficiency virus infected);
* Subjects who underwent treatment of any type of cancer within the last six months;
* Subjects with any pacemakers, or any metallic implants or prostheses in the vicinity of the treatment site (such as ankle, foot, etc.);
* Subjects with any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with study evaluations or optimal participation in the study;
* Subjects who may be unreliable for the study including Subjects who engage in excessive alcohol intake or drug abuse (no testing required), or Subjects who are unable to return for scheduled follow-up visits;
* Subjects who feel they cannot sit for 45 minutes at a time during the treatment.
* Subjects who are part of the staff personnel directly involved with this study;
* Subjects who are family members of the investigational study staff;
* Subjects with a history or signs of peripheral circulatory insufficiency and/or diabetic neuropathy;
* Subjects with known allergy to any of the tested treatment products [i.e. perfluorocarbons and plastic polycarbonate];
* Women who are pregnant, breastfeeding, or planning pregnancy prior to the end of study participation;

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey N Roe, PhD, Principal Investigator — DeviceFarm, Inc.
Locations (2):
- United States (2):
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Center For Clinical Research Inc., San Francisco, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Multi-center Open Label: 26 Subjects with 20-75% Distal Subungual Onychomycosis (mild to moderate DSO) infection of their big toe (hallux) nail infected by the dermatophytes Trichophyton (T.) rubrum or T. mentagrophytes will be enrolled. All Subjects will receive three 45-minute plasma treatments performed over a week.
  RenewalNail™ Plasma Treatment System: application of cold atmospheric plasma to a fungal infected toenail
Period: Overall Study
Arm/Group | Multi-center Open Label
Started | 26
Completed | 24
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Multi-center Open Label
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 57 [24 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 26
Positive KOH and fungal culture for T. rubrum or T. mentagrophytes [Count of Participants; unit: Participants] | 26

OUTCOME MEASURES:

1. Primary Outcome: Mycological Cure
Description: mycological cure defined as two consecutive negative cultures per FDA guideline
Time Frame: 2 cultures taken a week apart within 2 weeks after the first treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Multi-center Open Label
Number analyzed (Participants) | 24
Participants | 12

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Multi-center Open Label
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 6/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multi-center Open Label (N=26)
Staphylococcal infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multi-center Open Label (N=26)
erythema (Skin and subcutaneous tissue disorders) | 5 (5)
edema (Skin and subcutaneous tissue disorders) | 4 (4)
exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT03072550/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT03072550/SAP_001.pdf